CLINICAL TRIAL: NCT01740544
Title: Computerised Assessment of Visual Neglect Symptoms in Peripersonal Space
Acronym: KMS-Neglect 2
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Median Klinik Berlin-Kladow (Unknown); NeuroCure Clinical Research Center, Charite, Berlin (Other); Center for Stroke Research Berlin (Other); Free University of Berlin (Other); Humboldt-Universität zu Berlin (Other)
Responsible Party: Principal Investigator, Andreas Meisel, Prof. Dr. med. Andreas Meisel, Charite University, Berlin, Germany
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: KMS-Neglect 2
Record Dates: First submitted 2012-07-27; First posted 2012-12-04 (Estimated); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Visual Neglect
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cathodal tDCS in young study participants (Experimental): Cathodal tDCS in young study participants
  Interventions: Other: Cathodal tDCS
- Cathodal tDCS in elderly study participants (Experimental): Cathodal tDCS in elderly study participants
  Interventions: Other: Cathodal tDCS
- Sham tDCS in young study participants (Sham Comparator): Sham tDCS in young study participants
  Interventions: Other: Sham tDCS
- Sham tDCS in elderly study participants (Sham Comparator): Sham tDCS in elderly study participants
  Interventions: Other: Sham tDCS

INTERVENTIONS:
Other: Cathodal tDCS — Cathodal tDCS applied over the right PPC
  Arms: Cathodal tDCS in elderly study participants; Cathodal tDCS in young study participants
Other: Sham tDCS — Sham tDCS applied over the right PPC
  Arms: Sham tDCS in elderly study participants; Sham tDCS in young study participants

SUMMARY:
Healthy subjects will undergo cathodal stimulation of the right posterior parietal Cortex (PPC) and assessment of neglect-like symptoms in the encircling monitor system (EMS) as well as in a standard clinical test (Test Battery for Attention Performance, TAP, Zimmermann & Fimm, 1993). The aim of this study is to investigate whether cathodal stimulation leads to poorer test performance.

ELIGIBILITY:
Inclusion Criteria:

* Younger subjects

  * aged between 18 and 35 years
  * ability to provide written informed consent
  * right-handedness
* Elderly subjects

  * aged between 50 and 85 years
  * ability to provide written informed consent
  * right-handedness

Exclusion Criteria:

- Exclusion criteria for both groups:

* serious psychiatric disorders (including depression, psychosis) in the past
* severe neurological disorders (such as epilepsy, dementia, stroke) in the past
* current severe medical disorder
* drugs, medication or alcohol abuse at the time of the study
* severe traumatic brain injury or tumor in the past
* operations on the brain, trepanations
* metallic implants in the head / neck area (except in the mouth), such as screws, splinter, artificial cochlea, electrodes
* severe skin diseases (like eczema) or very sensitive skin in the head region in the past
* epilepsy in the family
* current use of neuroleptics, antiepileptics, antidepressants, L-dopa, benzo-diazepines
* current pregnancy or lactation
* current claustrophobia

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Test performance of young study participants in the encircling monitor system with/without cathodal stimulation
  Comparison of the young subjects' performance with vs. without transcranial direct current stimulation (tDCS) in the following computerised tests: Star Cancellation (number of omissions, latency & crossing index; based on Rabufetti, 2012), Landmark (reaction times, accuracy; based on Giglia et al., 2011), Visual Detection (reaction times, omissions; based on Sparing et al., 2009), Extinction (number of correct responses; based on Niedeggen & Hoffmann, 2011)

SECONDARY OUTCOMES:
Test performance of elderly study participants in the encircling monitor system with/without cathodal stimulation
  Comparison of the performance with vs. without transcranial direct current stimulation (tDCS) in the following tests: Star Cancellation, Landmark, Visual Detection, Extinction (see above)
Test performance of study participants in the Test Battery for Attention Performance (TAP) with/without cathodal stimulation
  Comparison of reaction times and number of omissions in the left and right visual field in the TAP subtest "Neglect" with vs. without tDCS.
Comparison of visual search patterns between neglect patients and healthy subjects with cathodal stimulation
  Comparison of visual search direction, structuredness (crossing index), and omissions in the Star Cancellation Test

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Meisel, MD, Principal Investigator — Charite - Universitätsmedizin Berlin (NeuroCure Clinical Research Center)
Locations (1):
- Charité University Medicine, Berlin, Germany